CLINICAL TRIAL: NCT04501835
Title: Assessment of Diagnostic and Therapeutic Practices for Cardiac Implantable Electronic Devices Suspected Infections in Nancy University Hospital
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PI077
Record Dates: First submitted 2020-07-20; First posted 2020-08-06 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2020-05

CONDITIONS: Cardiac Implantable Electronic Device Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac implantable electronic device infections: Patients hospitalised in Nancy University Hospital for suspected cardiac implantable electronic device infections
  Interventions: Other: Diagnostic and treatment evaluation

INTERVENTIONS:
Other: Diagnostic and treatment evaluation — No intervention, description of the diagnostic evaluation and the treatment

SUMMARY:
The frequency of cardiac implantable electronic devices (CIED) is constantly increasing.

Devices infections are one of the most serious complications in terms of morbidity and mortality. Although the frequency of cardiac implantable devices infections is difficult to derminate due to divergent definitions, cohort studies report a trend of increasing.

The infection can be localized at the pocket of the implantation, at intravascular or intra-cardiac portion of leads. Infectious endocarditis defined by involvement of the intra-cardiac portion of leads is the most serious form. The diagnosis is based on clinical, biological and multimodal imagery data. Early diagnosis and specific management are necessary to reduce mortality and morbidity.

Since the last European recommendations on infectious endocarditis in 2015, the HeartRythm Society of patient described an algorithm to treat CIED infections and extraction indications.

However, in practice, management of CEID infections remains center-dependent and data from robust international studies are missing.

The main objective of our study is to evaluate the management of CEID suspected infections and the prognosis at 1 year in terms of survival according to the methods of treatment at the Nancy University Hospital and to compare the treatment with the latest recommendations in force

ELIGIBILITY:
Inclusion Criteria:

* All patients who have been hospitalized in Nancy University Hospital between January 2014 et July 2019 for suspected infection of cardiac implantable electronic device

Exclusion Criteria:

* Minor patients
* Epicardial CIED

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in Nancy University Hospital between January 2014 et July 2019 for CIED suspected infection
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Description of the practice | From January 2014 to July 2020
  Describe the diagnostic and therapeutic practices of patients hospitalized for CIED suspected infection

SECONDARY OUTCOMES:
Evaluation of local practices against current recommendations | From January 2014 to July 2020
  * Classify patients in 3 groups (1 = Cardiac implantable electronic device infection ; 2 Pocket infection without proof of lead involvements ; 3 = systemic infection related to infective valvular endocarditis or not without proof of lead involvements according to our local practices and criteria, to EHRA criteria and modified Duke Li criteria).
  * Compare diagnostic management in our center with EHRA recommendations in each groups
  * Compare therapeutic management including removal/extraction of cardiac implantable electronic device, antibiotic therapy
  * Assessment of adhering to EHRA recommendations
  * Pronostic evaluation according to removal/extraction or not based on survival curve

CONTACTS AND LOCATIONS:
Locations (1):
- De Ciancio, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: Yes
Anonymous individual datas for baseline characteristcs and clinical outcomes would be available
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 1 year
Access Criteria: Data access request will be reviewed by investigator team. Requestors will be required to signe a data access agreement

REFERENCES:
- [Background] Greenspon AJ, Patel JD, Lau E, Ochoa JA, Frisch DR, Ho RT, Pavri BB, Kurtz SM. 16-year trends in the infection burden for pacemakers and implantable cardioverter-defibrillators in the United States 1993 to 2008. J Am Coll Cardiol. 2011 Aug 30;58(10):1001-6. doi: 10.1016/j.jacc.2011.04.033. PMID 21867833
- [Background] Joy PS, Kumar G, Poole JE, London B, Olshansky B. Cardiac implantable electronic device infections: Who is at greatest risk? Heart Rhythm. 2017 Jun;14(6):839-845. doi: 10.1016/j.hrthm.2017.03.019. Epub 2017 Mar 16. PMID 28315744
- [Background] Habib G, Lancellotti P, Antunes MJ, Bongiorni MG, Casalta JP, Del Zotti F, Dulgheru R, El Khoury G, Erba PA, Iung B, Miro JM, Mulder BJ, Plonska-Gosciniak E, Price S, Roos-Hesselink J, Snygg-Martin U, Thuny F, Tornos Mas P, Vilacosta I, Zamorano JL; ESC Scientific Document Group. 2015 ESC Guidelines for the management of infective endocarditis: The Task Force for the Management of Infective Endocarditis of the European Society of Cardiology (ESC). Endorsed by: European Association for Cardio-Thoracic Surgery (EACTS), the European Association of Nuclear Medicine (EANM). Eur Heart J. 2015 Nov 21;36(44):3075-3128. doi: 10.1093/eurheartj/ehv319. Epub 2015 Aug 29. No abstract available. PMID 26320109
- [Background] Kusumoto FM, Schoenfeld MH, Wilkoff BL, Berul CI, Birgersdotter-Green UM, Carrillo R, Cha YM, Clancy J, Deharo JC, Ellenbogen KA, Exner D, Hussein AA, Kennergren C, Krahn A, Lee R, Love CJ, Madden RA, Mazzetti HA, Moore JC, Parsonnet J, Patton KK, Rozner MA, Selzman KA, Shoda M, Srivathsan K, Strathmore NF, Swerdlow CD, Tompkins C, Wazni O. 2017 HRS expert consensus statement on cardiovascular implantable electronic device lead management and extraction. Heart Rhythm. 2017 Dec;14(12):e503-e551. doi: 10.1016/j.hrthm.2017.09.001. Epub 2017 Sep 15. No abstract available. PMID 28919379